CLINICAL TRIAL: NCT05602883
Title: The Effect of Music Therapy on Risk Perception and Sleep Quality in Preterm Birth Threat
Brief Title: Music Therapy in the Threat of Premature Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, yasemin hamlacı başkaya, Head of Midwifery Depatment, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29092022
Record Dates: First submitted 2022-09-29; First posted 2022-11-02 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Sleep Quality; Premature Labor; Risk-Taking
Keywords: premature birth threat; sleep quality; risk perception
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Obstetric Labor, Premature; Risk-Taking | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: While the experimental group will listen to music at night, Routine midwifery care will be applied to the control group.
Masking Description: Since there is no placebo group, masking will not be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental: Experimental group Pregnant women in this group will listen to a music of their choice for 30 minutes before going to bed at night.
  Interventions: Behavioral: music therapy
- Control group (No Intervention): Women in the control group will not be interfered with and will be followed in line with the routine follow-up protocol of the clinic.

INTERVENTIONS:
Behavioral: music therapy — Music is played for 30 minutes to the pregnant woman who is hospitalized due to the threat of premature birth.
  Arms: Experimental group

SUMMARY:
The scope of the study covers the effects of music therapy on risk perception levels and sleep quality in pregnant women hospitalized due to the diagnosis of premature birth threat.

DETAILED DESCRIPTION:
Premature labor is an action accompanied by cervical effacement and dilatation with contractions that occur between the 20th and 37th weeks of pregnancy, occur 2 times in 10 minutes or 3-4 times in 30 minutes, and last at least 30 seconds. The threat of premature birth is 20-37. It is a condition in which uterine contractions are not accompanied by cervical effacement and dilatation between weeks of pregnancy. Premature birth is one of the main causes of perinatal mortality and morbidity.

Although the prevalence of threat of premature birth differs from society to society, it was determined as 17.3% in our country. There is no definitive cure for threat of premature birth. Measures and treatments are applied to reduce the risk of preterm birth. These are classified as bed rest, sedation, hydration and tocolytic agents. In addition, pregnant women should be kept under surveillance and followed in the hospital for the correct diagnosis and management of treatment. Being sick and being hospitalized affect the pregnant woman's life in various ways; It increases anxiety and can disrupt life balance. In high-risk pregnancies, the stress experienced due to maternal or fetal problems is higher than in normal pregnancies. Experiencing intense stress during pregnancy causes suppression of the immune system, decreased fetal birth weight and increased risk of preterm birth. Being aware of the stressors and using appropriate stress coping methods in high-risk pregnancy may provide better health outcomes for the mother and baby.

Relaxation exercises, breathing exercises, physical exercise, dreaming (catathymia), yoga, massage therapy, acupuncture, biological feedback, providing social support, music therapy, strengthening spirituality are effective coping methods in coping with the stress that occurs in high-risk pregnancy. Music, which is one of these methods, is frequently used by health professionals. Music therapy causes the release of endorphins and provides relaxation in the muscles, lowers blood pressure, decreases heart rate and respiratory rate, and positively affects the emotional state, improves maternal condition and creates a comfortable environment for the fetus. There are studies showing that music reduces anxiety, stress and pain during preterm labor, delivery and cesarean section. It is also an inexpensive, safe, and easy-to-learn method by health care professionals. In a study by Yang et al. (2009), the effect of music therapy in reducing anxiety for women on antepartum bed rest was investigated. It was determined that anxiety levels and physiological responses during bed rest in the intervention group were significantly reduced by music therapy. It was concluded that music can be a cheap and effective method to reduce anxiety in high-risk pregnancies. In the study of Liu et al. (2010) on music, it was determined that music can be used as a non-medical coping method in reducing labor pain and anxiety. Health professionals should encourage pregnant women to listen to relaxing music, determine the appropriate time for listening to music (while doing daily chores, listening to a relaxing and pleasant music while taking a warm shower, etc.), providing comfort and giving attention to music. One of the important factors in ensuring the comfort of pregnant women in the hospital is sleep. Sleep quality has been strongly associated with a person's quality of life. Sleep disturbance in pregnant women has also been associated with an increase in inflammatory and oxidative stress markers that indicate endothelial damage and metabolic status.

Changes in sleep quality are closely related to stress and anxiety. However, music therapy, which is one of the inexpensive, easily applicable and accessible, non-pharmacological coping methods, has not been studied in pregnant women diagnosed with premature birth threat. Therefore, the aim of this study is to determine the effect of music therapy on risk perception and sleep quality in pregnant women diagnosed with preterm birth threat.

ELIGIBILITY:
Inclusion Criteria:

* Being hospitalized with a diagnosis of premature birth threat,
* be able to speak Turkish,
* be able to communicate verbally and in writing,
* volunteering to participate in research
* single pregnancy,
* be between 18-45 years old

Exclusion Criteria:

* be deaf,
* using sleep-related medication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Richard Campbell Sleep Quality Scale | 4 days
  The Richard Campbell Sleep Quality Scale is a 6-item scale that evaluates the depth of night sleep, the time to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep. The total score of the scale is evaluated over 5 items, and the 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation. As the score of the scale increases, the sleep quality of the patients also increases.
Risk Perception Scale in Pregnancy | 4 days
  The scale is a visual analog measuring tool. Just below each item on the scale is a 0-100 mm linear line with the words "no risk" and "extremely high risk". The total score of the scale; It is calculated by adding the scores for each of the nine items and dividing the obtained score by 9. The scale has no breakpoints. An increase in the score obtained from the scale is interpreted as an increase in the risk perception of the pregnant woman and her baby.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Hamlacı Baskaya, Study Director — Sakarya University
Locations (1):
- Zeynep Kamil Gynecology and Pediatrics Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu YH, Lee CS, Yu CH, Chen CH. Effects of music listening on stress, anxiety, and sleep quality for sleep-disturbed pregnant women. Women Health. 2016;56(3):296-311. doi: 10.1080/03630242.2015.1088116. Epub 2015 Sep 11. PMID 26361642
- [Result] Heaman MI, Gupton AL. Psychometric testing of the Perception of Pregnancy Risk Questionnaire. Res Nurs Health. 2009 Oct;32(5):493-503. doi: 10.1002/nur.20342. PMID 19606451
- [Result] Hansen IP, Langhorn L, Dreyer P. Effects of music during daytime rest in the intensive care unit. Nurs Crit Care. 2018 Jul;23(4):207-213. doi: 10.1111/nicc.12324. Epub 2017 Nov 20. PMID 29159864
- [Result] Nour NM. Premature delivery and the millennium development goal. Rev Obstet Gynecol. 2012;5(2):100-5. PMID 22866189
- [Result] Shin HS, Kim JH. Music Therapy on Anxiety, Stress and Maternal-fetal Attachment in Pregnant Women During Transvaginal Ultrasound. Asian Nurs Res (Korean Soc Nurs Sci). 2011 Mar;5(1):19-27. doi: 10.1016/S1976-1317(11)60010-8. Epub 2011 Apr 5. PMID 25029946
- [Result] Yang M, Li L, Zhu H, Alexander IM, Liu S, Zhou W, Ren X. Music therapy to relieve anxiety in pregnant women on bedrest: a randomized, controlled trial. MCN Am J Matern Child Nurs. 2009 Sep-Oct;34(5):316-23. doi: 10.1097/01.NMC.0000360425.52228.95. PMID 19713801
- [Result] Liu YH, Chang MY, Chen CH. Effects of music therapy on labour pain and anxiety in Taiwanese first-time mothers. J Clin Nurs. 2010 Apr;19(7-8):1065-72. doi: 10.1111/j.1365-2702.2009.03028.x. PMID 20492051